CLINICAL TRIAL: NCT00001467
Title: Genetic Analysis of Immune Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950066; 95-I-0066
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-08-21

CONDITIONS: DOK 8; STAT1; GATA2; Immunodeficiency; STAT3
Keywords: Primary Immunodeficiency Disorders; Immunologic Disorders; Mutation; Genetic Analysis; Natural History
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Primary Immunodeficiency Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blood relatives: blood related family members of proband
- Proband: person initially ill/studied/diagnosed

SUMMARY:
The purposes of this study are to 1) identify the genes responsible for certain immune disorders, 2) learn about the medical problems they cause, and 3) learn how to predict who is likely to develop these disorders and what the risk is of passing them on to children. The immune system is the body s defense system. Some immune deficiencies impair a person s ability to fight infections; others render a person susceptible to allergies, or to autoimmune diseases such as lupus or arthritis, in which the immune cells (white blood cells) attack and destroy the body s own tissues.

Patients with immune disorders known or suspected to have a genetic basis and their family members may enroll in this study. Eligibility will be determined by a review of the patient s medical records and family medical history. Participants will provide a small blood sample for genetic (DNA) and white blood cell analysis. Gene samples (but not white blood cells) may also be obtained by mouth brushing or skin biopsy. For the mouth brushing, a small brush is rubbed against the inside of the cheeks for 1 minute to wipe off some cells. For the skin biopsy, a small circle of skin (about 1/8 inch) is removed under local anesthetic. Pregnant women may be asked to provide a fetal sample (amniotic fluid cells or chorionic villus sample). All samples will be used for immune or genetic studies of the family s immune disorder.

If test results show a specific genetic variation responsible for the family s immune disorder, a report will be sent to the patient s doctor or genetic counselor, who will discuss the implications for the family. NIH researchers and genetic counselors will also be available to explain results and answer questions. Information will not be available in the case of disorders that cannot yet be linked to a specific genetic abnormality.

Information from this study will increase knowledge about the immune system and what causes immune deficiencies. Participants may also learn the underlying cause of an immune disorder that affects them or someone in their family information may be useful in guiding treatment and in making decisions regarding family planning.

DETAILED DESCRIPTION:
This protocol includes studies of genetic defects of the immune system that cause failure of host defenses against infections, immune dysregulation and autoimmune diseases. Numerous rare disorders result from inherited or newly arising mutations in genes involved in the development and function of innate and adaptive immune systems or both. As specific disease syndromes are defined and the responsible genes identified, mutations in individual families can be sought. Correlation of mutation sites with clinical information helps to determine how specific gene segments encode important functional domains of the proteins of the immune system within the same genetic defect. Rare, single gene disorders identify immunologic pathways that might contribute to more common conditions, such as failure to respond to vaccines, susceptibility to allergies, or autoimmune diseases like arthritis or lupus.

Members of families with immune disorders that are known or suspected to have a genetic basis may be eligible. Immunologic tests and DNA sequence analysis appropriate to each clinical condition will be performed as needed on affected individuals and at-risk family members. Healthy family members may serve as controls. Probands, parents of deceased affected individuals, or entire families, may be referred to the Investigators Initially, clinical and family history as well as laboratory data will be reviewed by the investigators to determine eligibility. Subjects considered appropriate will be invited through their referring physician to participate by signing our consent form and sending appropriate blood, DNA or other samples to our PI. Should a genetic basis for an individual s immune disorder be identified or if clinical eligibility for other protocols is met, they may be invited to visit NIH.

ELIGIBILITY:
* INCLUSION / EXCLUSION CRITERIA:

Probands and their blood relatives, of any age, and ethnicity, who are affected, or suspected of being affected with genetic conditions and immune dysregulations under study are eligible to enroll as patients and family member enrollees.

Ages: 1 Day to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Probands and their blood relatives, of any age, sex, and ethnicity, who are affected, or suspected of being affected with genetic conditions and immune dysregulations under study are eligible to enroll as patients or family member enrollees. Fetal samples may be studied in selected cases where benefit, such as expedited postnatal treatment, could be realized.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1995-06-06 (Actual)

PRIMARY OUTCOMES:
To search for modifiers of phenotype in subjects with disorders of the immune system in which penetrance and expressivity are variable. | blood draw and testing once or can be repeated
  Greater understanding of the variable penetrance and expressivity of modifiers of phenotype in subjects with disorders of the immune system
genetic testing for known or suspected mutations related to primary immune deficiencies | blood draw and testing once or can be repeated
  diagnosis of genetic mutations or deficiencies causing rare primary immune diseases under study

SECONDARY OUTCOMES:
To track the natural history of disease outcome in selected disorders. | over time via history and assignment to other protocols
  understanding of natural history of selected disorders
To perform genotype/phenotype analysis in subjects with immune defects of known genetic cause, leading to basic research on interactions between components of receptors in immune system pathways. | blood draw and testing once or can be repeated
  understanding of interactions between components of receptors in immune system pathways in immune defects of know genetic cause
To identify by clinical and laboratory studies, including mutation detection in patients and healthy relatives who may be carriers, subjects who may be eligible for related protocols or who may derive clinical benefit from molecular diagnosis. | upon known or suspected diagnosis
  To follow patients and relatives that are affected or carriers of genetic defects over time and gain of further understanding of the natural history of diseases/conditions of the immune system.caused by genetic mutations/deficiencies

CONTACTS AND LOCATIONS:
Overall Officials: Gulbu Uzel, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share human data generated in this study for future research as follows:@@@@@@-Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the NIH CC).@@@@@@-De-identified or identified data with approved outside collaborators under appropriate agreements.@@@@@@-Data sharing may be complicated or limited in certain cases by contractual obligations or agreements with outside collaborators, such as cooperative research and development agreements, clinical trial agreements, other restraints, etc.
Supporting Information: ICF
Time Frame: PD and supporting information will be available after completion of the study.
Access Criteria: Data will be shared through:@@@@@@-Approved outside collaborators under appropriate individual agreements.@@@@@@-Publication and/or public presentations.@@@@@@Data might be shared before publication.@@@@@@The PI will review all requests for sharing data.

REFERENCES:
- [Background] Puck JM. Molecular and genetic basis of X-linked immunodeficiency disorders. J Clin Immunol. 1994 Mar;14(2):81-9. doi: 10.1007/BF01541340. PMID 8195317
- [Background] Fisher GH, Rosenberg FJ, Straus SE, Dale JK, Middleton LA, Lin AY, Strober W, Lenardo MJ, Puck JM. Dominant interfering Fas gene mutations impair apoptosis in a human autoimmune lymphoproliferative syndrome. Cell. 1995 Jun 16;81(6):935-46. doi: 10.1016/0092-8674(95)90013-6. PMID 7540117
- [Background] Pepper AE, Buckley RH, Small TN, Puck JM. Two mutational hotspots in the interleukin-2 receptor gamma chain gene causing human X-linked severe combined immunodeficiency. Am J Hum Genet. 1995 Sep;57(3):564-71. PMID 7668284
- [Derived] Donko A, Sharapova SO, Kabat J, Ganesan S, Hauck FH, Bergerson JRE, Marois L, Abbott J, Moshous D, Williams KW, Campbell N, Martin PL, Lagresle-Peyrou C, Trojan T, Kuzmenko NB, Deordieva EA, Raykina EV, Abers MS, Abolhassani H, Barlogis V, Milla C, Hall G, Mousallem T, Church J, Kapoor N, Cros G, Chapdelaine H, Franco-Jarava C, Lopez-Lerma I, Miano M, Leiding JW, Klein C, Stasia MJ, Fischer A, Hsiao KC, Martelius T, Seppanen MRJ, Barmettler S, Walter J, Masmas TN, Mukhina AA, Falcone EL, Kracker S, Shcherbina A, Holland SM, Leto TL, Hsu AP. Clinical and functional spectrum of RAC2-related immunodeficiency. Blood. 2024 Apr 11;143(15):1476-1487. doi: 10.1182/blood.2023022098. PMID 38194689
- [Derived] West RR, Hsu AP, Holland SM, Cuellar-Rodriguez J, Hickstein DD. Acquired ASXL1 mutations are common in patients with inherited GATA2 mutations and correlate with myeloid transformation. Haematologica. 2014 Feb;99(2):276-81. doi: 10.3324/haematol.2013.090217. Epub 2013 Sep 27. PMID 24077845
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1995-I-0066.html